CLINICAL TRIAL: NCT02825342
Title: Proton Pump Inhibitor (PPI's) and Selective Serotonin Reuptake Inhibitor Therapy (SSRI's) for the Management of Non Cardiac Chest Pain (NCCP)
Brief Title: PPI's and SSRI's Therapy for the Management of NCCP
Acronym: NCCP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary endpoint was reached.
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Director, Evangelismos Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EvangelismosH
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Chest Pain Rule Out Myocardial Infarction
Keywords: Gastroesophageal Reflux Disease (GERD); Proton Pump Inhibitor (PPI)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Citalopram; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GERD with PPI's therapy (No Intervention): Patients will abnormal distal acid esophageal exposure will receive PPI twice daily for 8 weeks .
- PPI's and SSRI's therapy (Active Comparator): Patients with positive symptom index for chest pain will receive citalopram 20 mg once daily and PPI once daily for 8 weeks.
  Interventions: Drug: Citalopram
- SSRI's therapy (Active Comparator): Patients with a negative symptom index for chest pain will receive citalopram 20mg once daily for 8 weeks
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram
  Other Names: Proton Pump Inhibitor
  Arms: PPI's and SSRI's therapy; SSRI's therapy

SUMMARY:
Non cardiac chest pain (NCCP) is defined as recurring, angina-like, retrosternal chest pain of non cardiac origin. Annual prevalence of NCCP in the general population of the western world ranges from 25-35%. Of those patients presenting to an emergency room with chest pain, a cardiac etiology is ultimately found in only 11-39%. Several conditions are associated with NCCP, with gastroesophageal reflux disease (GERD) being the most prevalent, constituting up to 60% of cases. However, NCCP is considered a disorder of heterogenous nature and several other conditions, apart of GERD, such as esophageal dysmotility and esophageal hypersensitivity have been implicated.

Treatment of NCCP remains a real challenge due to the diverse underlying mechanisms responsible for patients' symptoms. Given the fact that GERD is by far the most common etiology, proton pump inhibitor (PPI) therapy has been tried extensively; however, after 6 weeks of treatment complete resolution of symptoms occurs in only 30% of patients, the optimal duration of PPI administration is not known, while the best maintenance dose has never been determined. Although the administration of selective serotonin reuptake inhibitors (SSRIs) could theoretically benefit those patients with esophageal hypersensitivity, the trials that have been published so far have included small number of patients and reported conflicting results, while the co-administration of PPIs with SSRIs has not been evaluated so far. Furthermore, data on treatment of patients with functional chest pain are lacking.

DETAILED DESCRIPTION:
We have therefore designed a prospective study in order to evaluate the effect of PPI and SSRI therapy for different subtypes of NCCP patients using multichannel intraluminal impedance and pH (MII-pH) monitoring.

METHODS

Patients with non cardiac chest pain symptoms presenting to the participating centres, will be prospectively screened for entry into the study.

They should have undergone a comprehensive diagnostic evaluation by cardiologists in order to exclude a cardiac source for their chest pain. Patients recruited in the study should have either a normal coronary angiogram or lack of ischemic heart disease on exercise treadmill or stress thallium testing

Inclusion criteria i) patients should have at least 3 episodes of chest pain per week in the previous 3 months.

The exclusion criteria will be:

i) thoracic, esophageal or gastric surgery ii) primary or secondary esophageal motility disorders iii) use of non-steroidal anti-inflammatory drugs and aspirin iv) presence of Barrett's esophagus, erosive esophagitis, peptic stricture and duodenal or gastric ulcer on upper endoscopy v) eosinophilic esophagitis vi) underlying psychiatric illness vii) pregnancy in women viii) refusal to participate.

Study protocol

All subjects who will agree to participate in the study should undergo an upper endoscopy to assess the presence or absence of esophageal mucosal injury. Patients with Barrett's esophagus and erosive esophagitis will not be included in the present study. Furthermore, biopsies will be taken and patients with eosinophilic esophagitis will also be excluded.

All patients will also be subjected to stationary esophageal manometry and those with motility abnormalities will be excluded. During esophageal manometry the lower esophageal sphincter (LES) will be located.

Esophageal impedance-pH monitoring will be performed in all participating subjects using an ambulatory multichannel intraluminal impedance (MII) and pH monitoring system (Sleuth; Sandhill Scientific, Inc. Higland Ranch, CO, USA). During the test, each subject will eat three standard meals, while the beginning and ending times of every meal will be indicated in a diary. Subjects will also be instructed to press the event marker button on the data logger whenever they experience chest pain. Data recording will be concluded after 24 hours, when patients will return to the endoscopy unit for the catheter removal.

The impedance and pH data will be used to determine in each patient the number and type of reflux episodes and the total 24-hour esophageal acid exposure, defined as the total time at pH below 4 divided by the time monitoring. Total distal esophageal acid exposure (i.e., % time pH < 4) less than 4.2% over 24 hours will be considered normal.

In each patient we will calculate the symptom index (SI) for chest pain. Bioview analysis software will be used for the calculation of SI. According to the setting of this software the symptoms will be considered as being related to reflux if they occur within a 2-min time window after the onset of the reflux episode. SI will be defined as the number of symptoms associated with reflux divided by the total number of symptoms. A positive SI is declared if ≥ 50% (i.e, at least half of the symptoms are associated with reflux).

Treatment

Patients will abnormal distal acid esophageal exposure will receive PPI twice daily for 8 weeks .

Patients with positive symptom index for chest pain will receive citalopram 20 mg once daily and PPI once daily for 8 weeks.

Patients with a negative symptom index for chest pain will receive citalopram 20mg once daily for 8 weeks.

All patients will be evaluated at the end of the 8-week period and will be asked about the presence or absence of chest pain. Treatment success will be defined as the complete disappearance of the chest pain, while the presence of mild or infrequent symptoms will be considered as treatment failure.

ELIGIBILITY:
Inclusion Criteria:

Patients should have at least 3 episodes of chest pain per week in the previous 3 months. Meanwhile they should have undergone a comprehensive diagnostic evaluation by cardiologists in order to exclude a cardiac source for their chest pain. Patients recruited in the study should have either a normal coronary angiogram or lack of ischemic heart disease on exercise treadmill or stress thallium testing.

Exclusion Criteria:

The exclusion criteria will be: i) a history of thoracic, esophageal or gastric surgery, ii) primary or secondary esophageal motility disorders, iii) use of non-steroidal anti-inflammatory drugs and aspirin, iv) presence of Barrett's esophagus, erosive esophagitis, peptic stricture and duodenal or gastric ulcer on upper endoscopy, v) eosinophilic esophagitis, vi) underlying psychiatric illness, vii) pregnancy in women, viii) refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
complete disappearance of the chest pain | at the end of the 8-week period of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No